CLINICAL TRIAL: NCT01611129
Title: Use of the 'Patient Journey' Model in the Internet-based Pre-fitting Counseling of a Person With Hearing Impairment: A Randomized Controlled Trial
Brief Title: Internet-based Pre-fitting Counseling of Persons With Hearing Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Lunner (Other Government)
Collaborators: Swansea University (Other)
Responsible Party: Sponsor-Investigator, Thomas Lunner, Professor, Linkoeping University
Organization: Linkoeping University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FAS-IT-03
Record Dates: First submitted 2012-05-14; First posted 2012-06-04 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Disability Evaluation
Keywords: Disability Evaluation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- reading about hearing loss and its management (Active Comparator): General self-reading reading about hearing loss and its management This would run for 30 days and the participants have to manage their own time.
  Interventions: Behavioral: Internet-based counseling
- Internet-based counseling (Experimental): This would involve 4 stages of designated internet sessions and additional tasks which the patients can complete in their own time. This programme should be completed within 30 days.
  Interventions: Behavioral: Internet-based counseling

INTERVENTIONS:
Behavioral: Internet-based counseling — Stage 1 - introduction to the concept of the patient journey and presenting the participants series of questions which may help them to explore their journey through hearing loss; Stage 2 - patient journey model of PHI and 2 case examples will be presented. The PHI will be advised to compare their journey to the model presented and identify the similarities and differences; Stage 3 - communication partners' journey model will be presented and the PHI will be asked to consider how interactions between each other may affect various things in the physical, mental and social domains; and Stage 4 - patients will be encouraged to think about how the PHI & CP may influence each other during their journey through hearing loss, how they can overcome some of the difficulties they may be experiencing and to think about the potential benefits and the challenges from the audiological management.

SUMMARY:
The purpose of this study is to determine whether the use of 'patient journey' model in internet-based counseling of a person with hearing impairment is a feasible approach in management of emotional and social consequences, anxiety and depression, readiness to change and acceptance of hearing loss.

ELIGIBILITY:
Inclusion Criteria:

* Ages over 18 years old
* Have symptoms of hearing difficulty
* Access to internet

Exclusion Criteria:

* HHQ results too low (i.e., below 20),
* Participants using hearing aids
* Those with additional disabilities (e.g., visual impairment, learning disability, dementia, and so on) which may affect individuals' ability to participate in an internet-based program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Hearing Handicap Questionnaire (HHQ) | One week pre-treatment, One week post treatment, Six-moths follow-up
  Change from baseline in reported emotional and social consequences due to hearing impairment one week post treatment.
  Hearing Handicap Questionnaire (HHQ) - Change from baseline

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | One week pre-treatment, One week post treatment, Six moths follow-up
  Change from baseline in reported depression and anxiety symptoms one week post treatment.
  Hospital Anxiety and Depression Scale (HADS) - Change from baseline
University of Rhode Island Change Assessment Scale (URICA) | One week pre-treatment, One week post treatment, Six months follow-up
  Change from baseline in readiness for change one week post treatment. University of Rhode Island Change Assessment Scale (URICA) - Change from baseline.
Hearing Impairment Acceptance Questionnaire (HIAQ) | One week pre-treatment, One week post treatment, Six months follow-up
  Change from baseline in acceptance of hearing loss one week post treatment. Hearing Impairment Acceptance Questionnaire (HIAQ) - Change from baseline.

CONTACTS AND LOCATIONS:
Locations (2):
- The Swedish Institute for Disability Research, Linköping University, Linköping, Sweden
- Department of Vision and Hearing Sciences, Anglia Ruskin University, Swansea, United Kingdom

REFERENCES:
- [Background] Manchaiah VK, Stephens D, Andersson G, Ronnberg J, Lunner T. Use of the 'patient journey' model in the internet-based pre-fitting counseling of a person with hearing disability: study protocol for a randomized controlled trial. Trials. 2013 Jan 24;14:25. doi: 10.1186/1745-6215-14-25. PMID 23347711
- [Derived] Manchaiah V, Ronnberg J, Andersson G, Lunner T. Use of the 'patient journey' model in the internet-based pre-fitting counseling of a person with hearing disability: lessons from a failed clinical trial. BMC Ear Nose Throat Disord. 2014 Apr 7;14(1):3. doi: 10.1186/1472-6815-14-3. PMID 24708677
- See also: Related Info — https://www.iterapi.se/sites/journey/